CLINICAL TRIAL: NCT01165918
Title: Basic Research. Unveiling Factors That Contribute to Germ Cell Differentiation
Brief Title: Derivation of New Human Embryonic Stem Cell Lines: Identification of Instructive Factors for Germ Cells Development
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Collaborators: Ben-Gurion University of the Negev (Other)
Responsible Party: Dr. Eitan Lunenfeld, Soroka Medical Center
Other Study IDs: Sor491210CTIL
Record Dates: First submitted 2010-07-06; First posted 2010-07-20 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-06

CONDITIONS: Normal Healthy Embryos

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Donated embryos

SUMMARY:
The purpose of this study is

1. To generate human embryonic stem cells lines (hESC) lines
2. Study of the factors that contribute to differentiation towards germ cell.

ELIGIBILITY:
Inclusion Criteria:

* any donated embryos

Exclusion Criteria:

* not relevant

Ages: 2 Days to 4 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: any donated embryo
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-10

PRIMARY OUTCOMES:
New hESC | 1 year
  Donated embryos will be used for derivation of the Es cells

SECONDARY OUTCOMES:
Factors that contribute to germ cells differentiation | 4 years
  We shall employ the knowledge from a study of sperm differentiation in mice to instruct the differentiation of ES cells towards germ cells

CONTACTS AND LOCATIONS:
Locations (1):
- Soroka medical center, Beersheba, Israel